CLINICAL TRIAL: NCT04802590
Title: A Randomized Phase II Trial Evaluating Ibrutinib Plus CD20 Ab and Venetoclax in Patients With Untreated Mantle Cell Lymphoma
Brief Title: Study of Ibrutinib + CD20 Antibody and Venetoclax in Patients With Untreated Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OASIS-II
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ibrutinib; venetoclax; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Ibrutinib (+ CD20Ab)
  Interventions: Drug: Ibrutinib 560 mg
- Arm B (Experimental): Ibrutinib + Venetoclax (+CD20Ab)
  Interventions: Drug: Ibrutinib 560 mg; Drug: Venetoclax 10 MG Oral Tablet [Venclexta]; Drug: Venetoclax 50 MG Oral Tablet [Venclexta]; Drug: Venetoclax 100 MG Oral Tablet [Venclexta]

INTERVENTIONS:
Drug: Ibrutinib 560 mg — 560mg/d continuously from C1D2 to end C24
Drug: Venetoclax 10 MG Oral Tablet [Venclexta] — 20mg/d from C2D1 to C2D7
  Arms: Arm B
Drug: Venetoclax 50 MG Oral Tablet [Venclexta] — 50mg/d from C2D8 to C2D14
  Arms: Arm B
Drug: Venetoclax 100 MG Oral Tablet [Venclexta] — 100mg/d from C2D15 to C2D21 200mg/d from C2D22 to C2D28 400mg/d from C3D1 to end C24
  Arms: Arm B

SUMMARY:
The OASIS II trial is a multicentre, open label, randomized phase II trial. We will compare the efficacy of Ibrutinib/anti-CD20 Ab versus Ibrutinib/anti-CD20 Ab/Venetoclax given as fixed duration combinations in newly diagnosed Mantle Cell Lymphoma (MCL) patients (≥ 18 years and < 80 years of age).

Treatment duration of Ibrutinib and Venetoclax will be a maximum of two years. Patients will be treated with CD20 Ab for 3.5 years.

The primary aim is to assess MRD status at 6 months in both arms.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years and < 80 years of age at the time of signing the informed consent form (ICF).
2. Patient understood and voluntarily signed and dated an ICF prior to any study-specific assessments/procedures being conducted.
3. Patient willing and able to adhere to the study visit schedule and other protocol requirements
4. Women of childbearing potential must have negative results for pregnancy test prior to study treatment start and agree to abstain from breastfeeding during study participation and at least 18 months after the last drug administration
5. Men or women of reproductive potential agree to use acceptable method of birth control during treatment and for eighteen months after the last drug administration.
6. Histologically confirmed (according to the World Health Organization (WHO) classification) mantle cell lymphoma. The diagnosis has to be confirmed by phenotypic expression of CD5, CD20 and cyclin D1 or the t(11;14) translocation (by cytogenetics and/or fluorescence in situ hybridization (FISH) and/or BCL1-IgH PCR)
7. Untreated MCL
8. Adequate renal function as demonstrated by a creatinine clearance > 50 mL/min; calculated by Cockcroft Gault formula or Modification of Diet in Renal Disease (MDRD)
9. Adequate hepatic function per local laboratory reference range as follow:

   * Aspartate transaminase (AST) and alanine transaminase (ALT) < 3.0 x upper limit of normal (ULN)
   * Bilirubin < 1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
10. Stage II-IV disease, measurable with at least lymph node > 1.5 cm and requiring treatment in the opinion of the treating clinician
11. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.
12. Life expectancy of more than 3 months.
13. For France: patient affiliated to any social security system

Exclusion Criteria:

1. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
2. Impaired organ function (other than liver and renal) which will interfere with the treatment
3. Hemoglobin level < 10g/dL; Neutrophil count <1 G/L; Platelets < 75 G/L (except if related to lymphoma then platelet must be >50),
4. Major surgery within 28 days before enrollment
5. Known central nervous system lymphoma
6. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
7. Requires anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon)
8. Requires treatment with strong CYP3A inhibitors
9. Vaccinated with live, attenuated vaccines within 6 months of enrollment (except COVID vaccine)
10. Known history of human immunodeficiency virus (HIV)
11. Evidence of other clinically significant uncontrolled condition(s) including but not limited to:

    * Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
    * Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. HBs antigen negative, anti-HBs antibody + and antiHBc antibody -) and subjects with anti-HB-core antibody that are HBV DNA negative may participate
12. Psychiatric illness or condition which could interfere with their ability to understand the requirements of the study
13. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator' opinion, could compromise the patient safety, interfere with the absorption or metabolism of treatment (Ibrutinib, CD20 Ab, venetoclax) or put the study outcomes at undue risk
14. Pregnant, planning to become pregnant, or lactating woman
15. Known hypersensitivity to study treatment (CD20 Ab, Ibrutinib, Venetoclax) or to any of the excipients
16. Known allergy to xanthine oxidase inhibitors or rasburicase
17. Known glucose-6-phosphate dehydrogenase (G6DP) deficiency
18. Known bleeding disorders
19. Severe prior reactions to monoclonal antibodies or with prior significant toxicity (other than thrombocytopenia) from Bcl-2 inhibitor
20. History of prior other malignancy with the exception of:

    * curatively treated basal cell carcinoma
    * curatively treated squamous cell carcinoma of the skin or carcinoma in situ of the cervix at any time prior to study
    * other curatively treated cancer and patient disease-free for over 5 years
21. Anti-cancer therapies including chemotherapy, radiotherapy or other investigational therapy, including targeted small molecule agents
22. Biological agents (e.g. monoclonal antibodies) for anti-neoplastic intent: excluded 30 days prior to first dose of venetoclax
23. Person deprived of his/her liberty by a judicial or administrative decision
24. Adult person under legal protection

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
Minimum residual disease (MRD) rate | 6 months
  Minimum residual disease rate using droplet digital PCR (ddPCR) in bone marrow (BM) and/or peripheral blood (PB) at the end of induction

SECONDARY OUTCOMES:
MRD rate | 6 months
  MRD response using quantified PCR (qPCR) in PB and BM
MRD rate | 12 months
  MRD response using ddPCR in PB and BM
MRD rate | 24 months
  MRD response using ddPCR in PB and BM
MRD rate | 3 months
  MRD response using ddPCR in PB
MRD rate | 18 months
  MRD response using ddPCR in PB
MRD rate | 30 months
  MRD response using ddPCR in PB
MRD rate | 36 months
  MRD response using ddPCR in PB
MRD rate | 42 months
  MRD response using ddPCR in PB
Overall response rate (ORR) | 3 months
  Overall response rate according to Lugano criteria
ORR | 6 months
  Overall response rate according to Lugano criteria
ORR | 12 months
  Overall response rate according to Lugano criteria
ORR | 18 months
  Overall response rate according to Lugano criteria
ORR | 24 months
  Overall response rate according to Lugano criteria
ORR | 30 months
  Overall response rate according to Lugano criteria
ORR | 36 months
  Overall response rate according to Lugano criteria
ORR | 42 months
  Overall response rate according to Lugano criteria
Complete response rate (CRR) | 3 months
  Complete response rate according to Lugano criteria
CRR | 6 months
  Complete response rate according to Lugano criteria
CRR | 12 months
  Complete response rate according to Lugano criteria
CRR | 18 months
  Complete response rate according to Lugano criteria
CRR | 24 months
  Complete response rate according to Lugano criteria
CRR | 30 months
  Complete response rate according to Lugano criteria
CRR | 36 months
  Complete response rate according to Lugano criteria
CRR | 42 months
  Complete response rate according to Lugano criteria
Progression free survival (PFS) | 5,5 years
  Progression free survival: time from randomization into the study to the first observation of documented clinical disease progression or death due to any cause
Overall survival (OS) | 5,5 years
  Overall survival from the date of randomization to the date of death from any cause
Duration of MRD negativity | 5,5 years
  time from the date of attainment the first negative MRD to the date of positive MRD
Delay from MRD positivity to clinical relapse | 5,5 years
  time from the date of attainment the first positive MRD based on PB or BM to the first observation of documented disease progression or death due to any cause
Duration of response | 5,5 years
  time from attainment of Complete Response (CR) or Partial Response (PR) to the date of first documented disease progression, relapse or death from any cause
Disease free survival | 5,5 years
  time from attainment of CR to the date of the first documented disease progression, relapse or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Steven Le Gouill, Principal Investigator — Lymphoma Study Association; Toby Eyre, Principal Investigator — NCRI UK; David Lewis, Principal Investigator — NCRI UK
Locations (45):
- Belgium (5):
  - A.Z. Sint Jan AV, Bruges
  - Universite Libre de Bruxelles - Hopital ERASME, Brussels
  - Hopital Jolimont, Haine-Saint-Paul
  - CHU de Liege, Liège
  - Universite Catholique de Louvain Mont Godinne, Yvoir
- France (35):
  - CHU d'Angers, Angers
  - CH d'Avignon - Hopital Henri Duffaut, Avignon
  - CH de la Côte Basque, Bayonne
  - CHU Jean Minioz, Besançon
  - Chu Morvan, Brest
  - Institut d'Hématologie de Basse Normandie, Caen
  - Chu Estaing, Clermont-Ferrand
  - CH Henri Mondor, Créteil
  - CHU de DIJON, Dijon
  - CHD de Vendée, La Roche-sur-Yon
  - CHU de Grenoble, La Tronche
  - CHRU de Lille, Lille
  - Hopital DUPUYTREN, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - Hopital St-Louis, Paris
  - Hopital NECKER, Paris
  - Chu de Bordeaux - Hopital Haut-Leveque - Centre Francois Magendie, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital de la Milétrie, Poitiers
  - Ch Annecy Gennevois, Pringy
  - CH de Cornouaille, Quimper
  - CHU de REIMS, Reims
  - CHU Pontchaillou, Rennes
  - Centre Henri BECQUEREL, Rouen
  - Hopital René Huguenin, Saint-Cloud
  - Institut de Cancérologie de la Loire Lucien Neuwirth, Saint-Priest-en-Jarez
  - Institut de Cancérologie Strasbourg Europe, Strasbourg
  - IUCT Oncopole, Toulouse
  - CHU Bretonneau, Tours
  - CHU Nancy Brabois, Vandœuvre-lès-Nancy
  - CH de Bretagne Atlantique - Hopital CHUBERT, Vannes
  - Institut Gustave ROUSSY, Villejuif
- United Kingdom (5):
  - The Christie NHS Foundation Trust, Manchester
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Royal Cornwall Hospital Trust, Truro

IPD SHARING:
Plan to Share IPD: No